CLINICAL TRIAL: NCT05898191
Title: Effect of Laser Therapy on Vaginal Tissue at Biomechanical, Histological and Molecular Level in Women With Pelvic Organ Prolapse - Pilot Study
Brief Title: Effect of Laser Therapy on Vaginal Tissue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute for the Care of Mother and Child, Prague, Czech Republic (Other)
Collaborators: Department of Obstetrics and Gynecology, Faculty of Medicine, CUNI, Pilsen, Czechia (Unknown); NTIS, Faculty of Applied Sciences, University of West Bohemia, Pilsen, Czechia (Unknown)
Responsible Party: Principal Investigator, Lucie Hympanova, Principal investigator, Institute for the Care of Mother and Child, Prague, Czech Republic
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UPMDPrague 07032019
Record Dates: First submitted 2023-04-05; First posted 2023-06-12 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Pelvic Floor Disorders; Vaginal Atrophy
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- laser (Experimental): laser treatment (Laser CO² MIXTO PRO, LASERING SRL, Modena, Italy; three sessions, one per month)
  Interventions: Other: vaginal laser treatment
- control (No Intervention): no intervention

INTERVENTIONS:
Other: vaginal laser treatment — non-ablative vaginal laser application
  Other Names: (Laser CO² MIXTO PRO, LASERING SRL, Modena, Italy)
  Arms: laser

SUMMARY:
Pelvic floor disorders, including prolapse, incontinence, and vulvovaginal atrophy decrease the quality of life of every fourth woman. Recent therapy including habits change, rehabilitation, surgery, or hormonal replacement is not possible in all patients. Laser therapy is currently being proposed as an alternative. Laser therapy was brought to the gynecological field from dermatology, where it is used for facial rejuvenation (wrinkles) and treatment of other skin abnormalities. In dermatology, the laser has proven its efficacy at the molecular and histological levels. However, this concept was brought to gynecology without comparable confirmation. The skin and vagina have a different structures, therefore effects of laser may differ. Patient satisfaction with the clinical effects of laser has been reported. However, based on recent reviews and sheep studies knowledge about histological and other effects is limited. The goal of this study is to gain knowledge about the histological, biomechanical effects and molecular effects of laser on vagina. Control samples were collected from women undergoing colporrhaphy. The laser group underwent laser treatment prior to the surgery. The gained knowledge may improve laser protocols and in the future maybe laser therapy will become standard treatment in urogynecology.

ELIGIBILITY:
Inclusion Criteria:

* pelvic organ prolapse stage II (cystocele Ba ≥ -1)
* planned surgical treatment (anterior colporrhaphy)
* menopausal

Exclusion Criteria:

* surgical treatment at a location of interest
* use of systemic or vaginal estrogens within last 12 months

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
uniaxial biomechanical analysis | within month after completion of specimens
  Young's modulus of elasticity at low and high deformations

SECONDARY OUTCOMES:
quantitative histological analysis - epithelial thickness | within 6 months after completion of specimens
  Hematoxylin-eosin - epithelial thickness (um)
quantitative immunohistochemistry -von Willebrand factor (vWF) | within 6 months after completion of specimens
  microvessels density (mm-2) The number of von Willebrand factor-positive microvessel profiles was divided by the sum of the areas of the counting frame and expressed as a two-dimensional density of microvessels (QA, quantity per area)
quantitative immunohistochemistry -orcein | within 6 months after completion of specimens
  elastin fibres - Area fraction ( %)
quantitative immunohistochemistry- picrosirius red | within 6 months after completion of specimens
  collagen I and III - Area fraction ( %)
molecular analysis - markers of inflammation | within 6 months after results of histological analysis
  PCR (polymerase chain reaction) - TGFB (Transforming growth factor beta)
molecular analysis - markers of inflammation | within 6 months after results of histological analysis
  PCR - IL- 1 (Interleukin-1)
molecular analysis - connective tissue remodeling | within 6 months after results of histological analysis
  PCR - COLL1 (collagen type I)
molecular analysis - connective tissue remodeling | within 6 months after results of histological analysis
  PCR - MMP 1 (Matrix Metallopeptidase 1)

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Hajkova Hympanova, MD, PhD, Principal Investigator — Institute for the Care of Mother and Child, Prague, Czech Republic
Locations (1):
- Institute for the care of mother and child, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] P. Gupta, M. J. Ehlert, and J. M. Bartley, "Diagnosis and Management of Complex Pelvic Floor Disorders in Women," vol. 22, no. 6, pp. 275-285, 2015.
- [Background] Cruz VL, Steiner ML, Pompei LM, Strufaldi R, Fonseca FLA, Santiago LHS, Wajsfeld T, Fernandes CE. Randomized, double-blind, placebo-controlled clinical trial for evaluating the efficacy of fractional CO2 laser compared with topical estriol in the treatment of vaginal atrophy in postmenopausal women. Menopause. 2018 Jan;25(1):21-28. doi: 10.1097/GME.0000000000000955. PMID 28763401
- [Background] Papadavid E, Katsambas A. Lasers for facial rejuvenation: a review. Int J Dermatol. 2003 Jun;42(6):480-7. doi: 10.1046/j.1365-4362.2003.01784.x. PMID 12786881
- [Background] Kauvar AN. Fractional nonablative laser resurfacing: is there a skin tightening effect? Dermatol Surg. 2014 Dec;40 Suppl 12:S157-63. doi: 10.1097/DSS.0000000000000200. PMID 25417568
- [Background] Reilly MJ, Cohen M, Hokugo A, Keller GS. Molecular effects of fractional carbon dioxide laser resurfacing on photodamaged human skin. Arch Facial Plast Surg. 2010 Sep-Oct;12(5):321-5. doi: 10.1001/archfacial.2010.38. PMID 20855774
- [Background] Conte C, Jauffret T, Vieillefosse S, Hermieu JF, Deffieux X. Laser procedure for female urinary stress incontinence: A review of the literature. Prog Urol. 2017 Dec;27(17):1076-1083. doi: 10.1016/j.purol.2017.09.003. Epub 2017 Oct 21. PMID 29033365
- [Background] Pitsouni E, Grigoriadis T, Falagas ME, Salvatore S, Athanasiou S. Laser therapy for the genitourinary syndrome of menopause. A systematic review and meta-analysis. Maturitas. 2017 Sep;103:78-88. doi: 10.1016/j.maturitas.2017.06.029. Epub 2017 Jun 27. PMID 28778337
- [Background] Hympanova L, Rynkevic R, Mori Da Cunha MGMC, Diedrich CM, Blacher S, De Landsheere L, Mackova K, Krofta L, Roovers JP, Deprest J. The ewe as an animal model of vaginal atrophy and vaginal Er:YAG laser application. Menopause. 2020 Nov 23;28(2):198-206. doi: 10.1097/GME.0000000000001679. PMID 33235032
- [Result] Nygaard I, Barber MD, Burgio KL, Kenton K, Meikle S, Schaffer J, Spino C, Whitehead WE, Wu J, Brody DJ; Pelvic Floor Disorders Network. Prevalence of symptomatic pelvic floor disorders in US women. JAMA. 2008 Sep 17;300(11):1311-6. doi: 10.1001/jama.300.11.1311. PMID 18799443